CLINICAL TRIAL: NCT03689608
Title: Daily vs Intermittent Restriction of Energy: Randomised Controlled Trial to Reduce Diabetes Risk (DIRECT)
Brief Title: Daily vs Intermittent Restriction of Energy: Controlled Trial to Reduce Diabetes Risk (DIRECT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Adelaide (Other)
Responsible Party: Principal Investigator, A/Prof Leonie Heilbronn, Associate Professor, University of Adelaide
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: R20180319
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Individuals at Risk of Developing Diabetes
Keywords: intermittent fasting; calorie restriction; overweight and obesity
MeSH Terms: conditions — Intermittent Fasting; Overweight; Obesity | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intermittent Fasting (IF) (Experimental): 3 days fasting per week
  Interventions: Other: Intermittent Fasting (IF)
- Daily Restriction (DR) (Experimental): daily energy restriction
  Interventions: Other: Daily Restriction (DR)
- standard care (SC) (Other): usual care
  Interventions: Other: standard care (SC)

INTERVENTIONS:
Other: Intermittent Fasting (IF) — Participants will fast 3 days per week. In fasting days, meal replacements at 30% of daily energy requirements will be provided for the first 6 months. Participants will have fortnightly nutrition assessment.
  Arms: Intermittent Fasting (IF)
Other: Daily Restriction (DR) — Participants are instructed to restrict energy intake by 30% of daily energy requirements. Meal replacements will be provided for the first 6 months. Participants will have fortnightly nutrition assessment.
  Arms: Daily Restriction (DR)
Other: standard care (SC) — Participants will receive current practice guidelines in a static information format, will not take part in any counselling or receive meal replacements.
  Arms: standard care (SC)

SUMMARY:
In this randomized controlled trial, the investigators will compare the long term effectiveness of intermittent fasting (IF) versus an energy matched moderate calorie restriction (CR) over 18 months, and relative to a non-active intervention standard control (SC) in individuals who are at increased risk of developing type 2 diabetes. All participants will be required to attend the blood tests following a 12-hour overnight fast for the "A" visit at Month 0, 2, 6 (active) and 18 (follow up).

Fast424hGlucose: A subset of 100 participants enrolled in either IF or CR group in the parent study will be fitted with a continuous glucose monitor (CGM) to measure 24-hour glycaemic profile at month 0 and month 6.

Fast4Switch: Additional bloods will be collected after a "B" visit at month 6 to compare the fed to fasted switch. The B samples will be collected after a 12-hour overnight fast (CR, SC) or 20-hour fast (IF) to assess the metabolic switch to fasting in metabolites and hormones.

Fast4Stress: Additional subcutaneous adipose tissue, urine and saliva samples will be collected in ~32 men in IF and CR groups at month 0 and 6 at A and B visits to examine changes in stress response and resistance markers.

Experience2Fast: In-depth, semi-structured interviews will be carried out at month-8 follow-up visit in a subset of completers from IF or CR groups to explore the experience of intervention diets and understand contributing factors towards change and maintenance of dietary behaviours.

Fast4Flux: Additional blood samples will be collected in ~100 individuals in SC, IF and CR groups at month 0, month 2 and month 6 at A visit to measure autophagic flux in peripheral blood mononuclear cells following treatment of whole blood.

ELIGIBILITY:
Inclusion Criteria:

* weight-stable (< 5 % fluctuation in their body weight for past 6-months at study entry)
* score 12 or greater on the AUSDRISK calculator
* HbA1c <48 mmol/mol (measured at screening)

Exclusion Criteria:

* Personal history/diagnosis (self-reported) of diabetes (type 1 or 2), major psychiatric disorders (schizophrenia, major depressive disorder, bipolar disorder, eating disorders), gastrointestinal disorders, haematological disorders (i.e. thalassemia, iron-deficiency anaemia) insomnia, or any other medical condition, deemed unstable by the study physician.
* Participants currently taking the following medications will be excluded from participating: any medication used to lower blood glucose or antidiabetic medications (metformin, sulfonylureas, Glucagon-like peptide-1 GLP-1 analogues [i.e. exenatide], thiazolidinediones or DPP-IV inhibitors [i.e. 'gliptins']), medications affecting weight, appetite or gut motility (i.e. domperidone, cisapride, orlistat, phentermine, topiramate). Participants who are taking stable doses (i.e. > 12 months) of androgenic medications (i.e. testosterone) or SSRI's will not be excluded.
* weight change in past 3 months (> 5% screening weight)
* uncontrolled asthma, current fever, upper respiratory infections
* individuals who regularly perform high intensity exercise (>2 week)
* current intake of > 140g alcohol/week
* current smokers of cigarettes/cigars/marijuana/e-cigarettes/vaporisers
* current intake of any recreational drugs
* regular blood donor
* unable to comprehend study protocol due to English language or cognitive difficulties

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose AUC | 6 months
  Change in postprandial glucose AUC

SECONDARY OUTCOMES:
HbA1c | 2 months, 6 months, 18 months
  Change in HbA1c
Postprandial glucose | 18 months
  Change in postprandial glucose
Body weight | 2 months, 6 months, 18 months
  Change in body weight in kilograms
Body composition | 6 months, 18 months
  Change in body fat mass (kg) and fat free mass (kg)
Waist and hip circumference | 2 months, 6 months, 18 months
  Change in waist and hip circumference
Blood lipids | 2 months, 6 months, 18 months
  Changes in blood lipid profile (total cholesterol, HDL-, LDL-cholesterol and triglycerides)
Dietary intake | 2 months, 6 months, 18 months
  Change in food intake measured by self-reported food diaries
Blood pressure | 2 months, 6 months, 18 months
  Change in systolic blood pressure and diastolic blood pressure (mmHg)
Changes in physical Activity assessed by accelerometer | 2 months, 6 months, 18 months
  Change in average step counts measured with waist-worn actigraphy monitors
Fasting glucose | 2 months, 6 months, 18 months
  Change in fasting glucose
Fasting insulin | 2 months, 6 months, 18 months
  Change in fasting insulin
Fasting non-esterified fatty acids (NEFA) | 2 months, 6 months, 18 months
  Change in fasting NEFA levels
Fasting triglyceride | 2 months, 6 months, 18 months
  Change in fasting triglyceride levels
Postprandial insulin | 6 months, 18 months
  Change in postprandial insulin
Postprandial non-esterified fatty acids (NEFA) | 6 months, 18 months
  Change in postprandial NEFA levels
Postprandial triglyceride | 6 months, 18 months
  Change in postprandial triglyceride levels

OTHER OUTCOMES:
Change in perceived hunger and fullness assessed by visual analogue scales (VAS) | 6 months, 18 months
  Change in subjective hunger and fullness ratings measured by 0-100 mm VAS scales
Change in perceived sleep quality | 2 months, 6 months, 18 months
  Change in perceived sleep quality assessed by Pittsburgh Sleep Quality Index (PSQI), with a range from 0-21 scores, higher score reflect poorer sleep quality
Change in perceived eating behaviour | 2 months, 6 months, 18 months
  Change in perceived eating behaviour assessed by Three Factor Eating Questionnaire (TFEQ), which consists of 51 items to assess dietary restraint (21 items), disinhibition (16 items) and hunger (14 items), higher scores reflect higher levels on each subscale
Change in perceived quality of life | 2 months, 6 months, 18 months
  Change in perceived quality of life assessed by 36-item Short Form (SF-36) health survey, with a range from 0-100 scores, higher scores reflect better quality of life
Change in perceived well-being | 2 months, 6 months, 18 months
  Change in perceived well-being assessed by Personal Well-being Index, with a range from 0-10 scores, higher scores reflect greater satisfication
Change in food addition score | 6 months, 18 months
  Change in self-reported food addiction assessed by Yale Food Addiction Score (YFAS), with a range from 0-7 scores, higher scores reflect greater food addiction symptoms
Change in psychological distress | 6 months, 18 months
  Change in self-reported psychological distress assessed by Kessler Psychological Distress Scale (K10) , with a range from 10-50 scores, higher scores reflect higher psychological distress
Change in self-reported depression, anxiety and stress level | 2 months, 6 months, 18 months
  Change in self-reported depression, anxiety and stress level assessed by Depression, Anxiety and Stress Scale (DASS), with a range from 0-42 scores on each subscale, higher scores reflect higher levels on each subscale
Change in self-reported mood | 2 months, 6 months, 18 months
  Change in self-reported mood assessed by Positive and Negative Affect Schedule (PANAS), with a range from 0-100 scores, higher scores reflect more positive mood and negative mood.
Change in glucagon-like peptide 1 (GLP-1) | 6 months
  Change in glucagon-like peptide 1 (GLP-1)
Change in peptide YY | 6 months
  Change in peptide YY
Change in ghrelin | 6 months
  Change in ghrelin
Change in gastric inhibitory polypeptide (GIP) | 6 months
  Change in gastric inhibitory polypeptide (GIP)
Change in estradiol | 6 months
  Change in estradiol
Change in testosterone | 6 months
  Change in testosterone
Change in glucose (DIRECT- Fast4Switch) | 6 months
  Change in glucose levels
Change in non-esterified fatty acids (DIRECT- Fast4Switch) | 6 months
  Change in non-esterified fatty acids levels (NEFA)
Change in insulin (DIRECT- Fast4Switch) | 6 months
  Change in insulin levels
Change in triglycerides (DIRECT- Fast4Switch) | 6 months
  Change in triglycerides levels
24 hours glycaemia (DIRECT-Fast424hGlucose) | 6 months
  Changes in 24 hours glycaemia assessed by continuous glucose monitor
Salivary cortisol (DIRECT-Fast4Stress) | 6 months
  Change in salivary cortisol
Gene expression (DIRECT- Fast4Stress) | 6 months
  Change in gene expression
Change in urinary adrenaline (DIRECT- Fast4Stress) | 6 months
  Change in urinary adrenaline
Change in urinary noradrenaline (DIRECT- Fast4Stress) | 6 months
  Change in urinary noradrenaline
Qualitative analysis (DIRECT-Experience2Fast) | 8 months
  Patterns of participant's behaviour, characteristics and motivation that assist in or hinder from weight loss achievement by semi-structured interviews
Change in autophagic flux (DIRECT-Fast4flux) | 2 months, 6 months
  Change in autophagic machinery protein LC3B-II in peripheral blood mononuclear cells following treatment of whole blood.

CONTACTS AND LOCATIONS:
Overall Officials: Leonie Heilbronn, PhD, Principal Investigator — The University of Adelaide
Locations (1):
- University of Adelaide, Adelaide, South Australia, Australia

REFERENCES:
- [Derived] Teong XT, Liu K, Vincent AD, Bensalem J, Liu B, Hattersley KJ, Zhao L, Feinle-Bisset C, Sargeant TJ, Wittert GA, Hutchison AT, Heilbronn LK. Intermittent fasting plus early time-restricted eating versus calorie restriction and standard care in adults at risk of type 2 diabetes: a randomized controlled trial. Nat Med. 2023 Apr;29(4):963-972. doi: 10.1038/s41591-023-02287-7. Epub 2023 Apr 6. PMID 37024596
- [Derived] Teong XT, Liu K, Hutchison AT, Liu B, Feinle-Bisset C, Wittert GA, Lange K, Vincent AD, Heilbronn LK. Rationale and protocol for a randomized controlled trial comparing daily calorie restriction versus intermittent fasting to improve glycaemia in individuals at increased risk of developing type 2 diabetes. Obes Res Clin Pract. 2020 Mar-Apr;14(2):176-183. doi: 10.1016/j.orcp.2020.01.005. Epub 2020 Feb 11. PMID 32057716

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT03689608/SAP_000.pdf